CLINICAL TRIAL: NCT05347927
Title: Exploratory, Prospective, Multicenter, Observational Study to Evaluate the Influence of Undercast Material Types on Skin Microbiome
Brief Title: Observational Study to Evaluate the Influence of Undercast Material Types on Skin Microbiome
Acronym: Microbiome II
Status: Completed | Type: Observational
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: C2753
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Skin Microbiome; Undercast Materials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin microbiome swabs are collected for micribiome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: will receive water resistante padding and a cast
  Interventions: Device: water resistante padding
- Control group: will receive traditional non-water resistante padding and cast
  Interventions: Device: non water resistante padding

INTERVENTIONS:
Device: water resistante padding — * Delta-Dry® Softliner
  * Tensoban®
  * Delta-Dry®
  Groups: Test group
Device: non water resistante padding — * Delta-Net® Stockinette
  * Delta-Rol®
  Groups: Control group

SUMMARY:
This clinical study will evaluate the clinical performance and the safety of the CE-marked casting and padding materials when used in routine fracture care without any additional invasive methods and within the intended use. As primary objective the cast therapy´s influence on skin microbiome during fracture management will be investigated. Further, the influence of the padding material on the skin microbiome, device comfort, skin conditions, and impact on daily life activities as well as HCP´s and patient´s satisfaction and general product safety and performance are considered as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years of age
2. Patient is physically and mentally able to participate in this study
3. Proper understanding of the Dutch language
4. Signed informed consent
5. Fractures to be treated with a short-arm cast without thumb inclusion for the period of 3 weeks (e.g. 2R3A1 = radial styloid avulsion, 2R3A2 = Simple radial fracture, 2U3A1 = Ulnar fracture of the base of the styloid process, 2U3A2= Simple distal ulna fracture, 2R3B1 = Intraarticular fracture of the styloid process of the radius (not displaced) or Triquetrum fracture (non AO classified))

Exclusion Criteria:

1. Subject <18 years of age
2. Pregnancy, breast feeding
3. Participation in other clinical trials
4. Patient is neither physically nor mentally able to participate in this study
5. Non-intact skin in treatment area (including dermatological issues)
6. Patients with impaired (e.g. Cortisone skin, extremely dry skin, parchment skin) or damaged skin with either a surgical wound or a traumatic wound
7. Medical treatment prior casting which could influence the microbiome
8. Known Blood Circulatory Diseases
9. Known Lymphedema or any general disorder of the lymphatic system
10. Known Osteoporosis
11. Known Diabetes
12. Knowing of one of the following illnesses that might require regular systemic medication: cancer, rheumatic disease
13. Intolerability or documented allergies against cast materials
14. Subjects with not "normal" (unusual) hygienic behavior
15. Suspected drug addiction or alcohol abuse
16. Patients diagnosed HIV-positive or with infectious hepatitis based on self-declaration by subjects

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with broken forwarm receiving short arm cast
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
products´ influence on skin microbiome during fracture management | 3 weeks
  Quantity of bacteria in the skin microbiome
products´ influence on skin microbiome during fracture management | 3 weeks
  Taxonomic composition of skin microbiome
products´ influence on skin microbiome during fracture management | 3 weeks
  Alpha diversity of skin microbiome
products´ influence on skin microbiome during fracture management | 3 weeks
  Beta diversity skin microbiome

SECONDARY OUTCOMES:
Number of adverse events during study per product | 3 weeks
General product performance | 3 weeks
Treatment comfort | 3 weeks
Impact on daily life activities | 3 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Ommelander Ziekenhuis, Groningen, Scheemda
  - Wilhelmina Ziekenhuis Assen (Assen, NL), Assen
  - Leids Universitair Medisch Centrum (Leiden, NL), Leiden

IPD SHARING:
Plan to Share IPD: No